CLINICAL TRIAL: NCT03281473
Title: Comparison of Positive End Expiratory Pressure Titration Methods in Patients With Acute Respiratory Distress Syndrome: a Physiological Study
Brief Title: Comparison of Positive End Expiratory Pressure Titration Methods in ARDS Patients
Acronym: ELSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 49RC17_0220
Record Dates: First submitted 2017-07-11; First posted 2017-09-13 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Esophageal pressure; Mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms A (Experimental): Strategy 1 - Washout period - Strategy 2
  Interventions: Other: Strategy 1; Other: Strategy 2
- Arms B (Experimental): Strategy 2 - Washout period - Strategy 1
  Interventions: Other: Strategy 1; Other: Strategy 2

INTERVENTIONS:
Other: Strategy 1 — PEEP titration according to transpulmonary-end-expiratory pressure
Other: Strategy 2 — PEEP titration according to chest wall elastance measurement

SUMMARY:
This study aims at assessing the short-term physiological effects of 2 positive end expiratory pressure titration strategies in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Moderate or severe ARDS
* Consent to participation obtained from a relative

Exclusion Criteria:

* Protect adult
* Pregnant or breastfeeding woman
* No-affiliation to the social security scheme
* Contra-indication to the placement of an esophageal pressure measuring catheter
* Pneumothorax
* Hemodynamic and / or respiratory instability
* Extra-corporeal membrane oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Short-term effects of 2 PEEP titration strategies on gas exchange | 2 hours 15 minutes

SECONDARY OUTCOMES:
Short-term effects of 2 PEEP titration strategies on respiratory mechanics | 2 hours 15 min
Short-term effects of 2 PEEP titration strategies on hemodynamics | 2 hours 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Study Official is required by the WHO and BELONCLE, Ass.Pr, Principal Investigator — Angers teatching hospital
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chean D, Courtais A, Pavlovsky B, Yvin E, Desprez C, Taillantou-Candau M, Piquilloud L, Richard JC, Mercat A, Beloncle FM. Comparison of two transpulmonary pressure-based positive end-expiratory pressure titration strategies in acute respiratory distress syndrome: a randomized crossover study. Crit Care. 2025 Sep 29;29(1):409. doi: 10.1186/s13054-025-05626-x. PMID 41024114